CLINICAL TRIAL: NCT04830423
Title: The Effectiveness of Ultrasound Guided Intraarticular and Periarticular Ozone (O2-O3) Injection in the Treatment of Patients With Knee Osteoarthritis
Brief Title: The Effectiveness of Ultrasound Guided Ozone (O2-O3) Injection With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sefa Gümrük Aslan, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-04

CONDITIONS: Knee Osteoarthritis
Keywords: ozone injection; steroid injection; ultrasound; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- medikal ozone group (Active Comparator): medical ozone group patients diagnosed with knee ostheoarthritis
  Interventions: Procedure: Medical ozone injection
- steroid group (Other): steroid group patients diagnosed with knee ostheoarthritis
  Interventions: Procedure: steroid injection group

INTERVENTIONS:
Procedure: Medical ozone injection — Patients in the ozone (O2-O3) injection group will be given intraarticular and periarticular knee injections 3 times as the first dose of 10 μg / ml, the second dose is 15 μg / ml, and the third dose is 20 μg / ml, each session in a volume of 10 ml. Patients will be evaluated according to the study criteria at the beginning, 4 and 12 weeks later by a blinded investigator.
  Arms: medikal ozone group
Procedure: steroid injection group — In the steroid injection group, 1 ml of betamethasone (6 mg / ml) will be injected once intraarticular knee injection. Patients will be evaluated according to the study criteria at the beginning, 4 and 12 weeks later by a blinded investigator.
  Arms: steroid group

SUMMARY:
Knee ostheoarthritis (KOA) is a common disabling and degenerative disease leading to painful joints, articular stiffness, and decreased function. The mechanism of the ozone of relieving the pain and improving the knee function is through inhibiting the inflammation reaction in the KOA directly. Actually, the ozone intra-articular injection had been used to relieve the pain caused by KOA.

The aim of this study is to evaluate the effect of intra-articular injection of medical ozone given into the knee of the osteoarthritis patients, and to compare it with intra-articular steroid injection and to investigate the effectiveness of ozone and steroid the job to determine the superiority of the injections to each other.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. 96 people who met the inclusion criteria were randomized into two groups of people. The first group will be designated as Ozone group will be applied to these patients. Patients in the second group will be designated as the steroid group, and injections will be applied in accordance with protocol. Participants were evaluated with Visual Analogue Scale (VAS), The Western Ontario and McMaster Universities Arthritis Index (WOMAC). The presence of suprapatellar effusion of the participants whose evaluations are completed will be evaluated by ultrasonography and the findings will be recorded. Initial evaluations of the participants will be made before the first injection. Patients in the ozone (O2-O3) injection group will be given intraarticular and per-articular knee injections 3 times as the first dose of 10 μg / ml, the second dose is 15 μg / ml, and the third dose is 20 μg / ml, each session in a volume of 10 ml. In the steroid injection group, 1 ml of betamethasone (6 mg / ml) will be injected once intraarticular knee injection. Patients will be evaluated according to the study criteria at the beginning, 4 and 12 weeks later by a blinded investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Female / male aged> 45 years
2. Diagnosis of knee ostheoarthritis after physical examination and imaging (direct radiography)
3. Those whose symptoms persist> 6 months
4. Radiological staging of osteoarthritis according to the Kellgren-Lawrence scale Grade 2 and 3
5. Participation in the study voluntarily and regularly

Exclusion Criteria:

1. History of previous knee surgery
2. Patients with inflammatory arthritis (Rheumatoid arthritis, psoriatic arthritis, gouty arthritis as)
3. Patients with neuropathic pain
4. Those with pain reflected from the waist or hip
5. History of tumor, infectious, psychiatric illness, bleeding diathesis
6. Trauma history within the last 6 months
7. Hyaluronic acid or steroid injection in the last 3 months
8. Those with systemic diseases such as diabetes, rheumatoid arthritis, hepatitis, coagulopathy
9. Those with malignant hypertension
10. Those with G6PDH (Glucose 6-Phosphate Dehydrogenase) deficiency
11. Those with Graves' disease
12. Those with cerebrovascular event disease in which bleeding continues actively

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
PAIN - Numerical Rating Scale (NRS) | up to 12 weeks
  Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Severity of pain was assessed NRS using the standard 10 cm (at rest, at motion and at night) with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end.

SECONDARY OUTCOMES:
Quality of life - Short Form-36 (SF-36) | initial, 4th week 12th week pain change
  Satisfaction assessed by the SF-36. Short Form (SF-36) was used to investigate the quality of life of the patients.The reliability and validity of the Turkishversion of SF-36 has been demonstrated. SF-36 consists of 36 questions on eight different subscales including physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, energy and fatigue, vitality, social functioning, role limitations due to emotional problems and general mental health. Each subscale of SF-36 is scored between 0 and 100, and higher scores show better Quality of life.
PAIN, PHYSICAL FUNCTION -Western Ontario and McMaster Universities Arthritis Index (WOMAC) | initial, 4th week 12th week pain change
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:Pain, Stiffness and Physical Function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Sefa Gümrük Aslan, Principal Investigator — Gaziler Physical Medicine And Rehabilitation Health Application And Research Center
Locations (1):
- Sefa, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No